CLINICAL TRIAL: NCT04216966
Title: Evaluation of Root Roughness and Smear Layer Formation Using Conventional and Contemporary Dental Curettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Collaborators: University of Karachi (Other)
Responsible Party: Principal Investigator, Sania Riaz, post graduate trainee, Dow University of Health Sciences
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 14071985
Record Dates: First submitted 2019-12-18; First posted 2020-01-03 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Dental Calculus
MeSH Terms: conditions — Dental Calculus | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The scanning electron photographs were assessed by assessors who were blinded to the study groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Placebo Comparator): This group did not undergo any instrumentation.
  Interventions: Device: Control group
- Gracey Curette group (Experimental): Teeth under this group were subjected to debridement with Gracey curette .
  Interventions: Device: Gracey Curette
- After Five group (Experimental): Teeth under this group were subjected to debridement with After 5 curette .
  Interventions: Device: After Five
- Mini Five group (Experimental): Teeth under this group were subjected to debridement with Mini Five curette .
  Interventions: Device: Mini Five

INTERVENTIONS:
Device: Control group — No intervention was given
  Arms: Control group
Device: Gracey Curette — Lingual surface of tooth was debrided by Gracey Rigid curette
  Other Names: 5/6 Gracey Rigid curette (Hu-Friedy Co, Chicago, IL, US)
  Arms: Gracey Curette group
Device: After Five — Lingual surface of tooth was debrided by After Five Rigid curette
  Other Names: 5/6 After Five Rigid curette (Hu-Friedy Co, Chicago, IL, US)
  Arms: After Five group
Device: Mini Five — Lingual surface of tooth was debrided by Mini Five Rigid curette
  Other Names: 5/6 Mini Five Rigid curette (Hu-Friedy Co, Chicago, IL, US)
  Arms: Mini Five group

SUMMARY:
The objective of the present study is to evaluate the surface texture of root after hand instrumentation with Gracey curette, After Five curette and Mini Five curette.Patients having chronic periodontitis and scheduled for extraction were randomized into four groups. Scaling and Root planing was performed by different curettes. Group 1 didn't under go any instrumentation. Group 2 was instrumented with Gracey curette, Group 3 with After Five curette and Group 4 with Mini Five curette. These hopeless teeth were then extracted atraumatically and the specimens were processed and analyzed under a Scanning Electron Microscope. "Roughness and Loss of Tooth substance index" and "Smear layer index" was evaluated using the Scanning Electron Microscope photographs.Means and frequencies were reported using SPSS Version-21.Cross Tabulation was made between the test groups (Control, Gracey Curette, After five and Mini Five) versus "Roughness and Loss of Tooth substance Index" and "Smear Layer Index". Chi square test was applied to see the grade distribution among groups. Frequencies were reported in percentages and means. P. value of 0.05 or less was considered as significant.

DETAILED DESCRIPTION:
INTRODUCTION:

The main objective of scaling and root planing is to smoothen the root surface.Scaling and root planing can be done with a variety of instruments, however, hand instruments are still considered the "gold standard" for treatment. Hand and ultrasonic instruments are primarily used for debridement and produces root surface irregularities which enhances colonization of bacteria, deposition of plaque and retain more calculus.It is also a known fact that these debridement procedures produce a smear layer on the root surface which is detrimental to the healing and regeneration of periodontal tissues, as it interferes with the reattachment of cells derived from the periodontal ligament to the root surface.16

Objective:

The objective of the present study is to evaluate the surface texture of root after hand instrumentation with Gracey curette, After Five curette and Mini Five curette.

Study Design:

A Single Blinded Randomized Control Trial

Study Setting:

The study was conducted in the Periodontology Department of Dr. Ishrat-ul-Ebad Khan Institute of Oral Health Sciences Sample Size Using PASS software version 11, two independent sample t-test, 95% confidence interval, 80% power of test, roughness mean and standard deviation in group 1,hand instrument (1.2 ± 0.3um)54 and group 2,control (1.1 ± 0.56um)54 calculated sample size was 99 which was raised upto 120 teeth.

Sampling Technique:

Consecutive sampling

Clinical Procedure:

120 patients with ages between 35 - 60 years, having severe chronic periodontitis and scheduled for extraction were selected for this study. Detailed history was taken and a consent form was signed by the patient. Lingual surface of each tooth were subjected to debridement with any one of the test curettes. Patients were randomly assigned to any one of the four groups. Randomization was done by computer generated randomizing method. Randomization chart is given at the back.

Subgingival Instrumentation was performed in vivo by a single operator by either 5/6 Gracey Rigid Curette, 5/6 After Five Rigid Gracey curette or 5/6 Mini Five Rigid Gracey Curette. One group was not instrumented and kept as control. Local Anesthesia was given and scaling and root planing was performed until a smooth hard surface was detected by Explorer number 17. Following instrumentation, a small diamond round bur on a high speed hand piece was used to mark the level of the free gingival margin, lingually. This groove provided a landmark for evaluation under scanning electron microscope.

Instrumentation was carried out in vivo by a single operator trained in Periodontology, by a standard protocol. Modified pen grasp technique was used for holding the curettes. The angle between the cutting edge of the curette and the teeth was around 80 degree along with a good finger rest hence permitting a proper wrist-forearm motion. The shank of the instrument was kept parallel to the long axis of tooth. Degree of sharpness was maintained by sharpening the curettes after every 5 strokes with Arkansas stone.( Hu-Friedy Co, Chicago, IL, US) .The tooth were then extracted atraumatically as possible, with the beak of extraction forceps above the gingival margin. After extraction the teeth were rinsed in running tap water for 60 seconds to remove all the debris and blood and placed in 0.9% NaCl solution for hydration until treatment.After instrumentation the samples were fixed in 2.5 % gluteraldehyde solution in phosphate buffer (pH 7.3) for 24 hours and then washed with phosphate buffer 3 times. All specimens were kept for 10 minutes in graded series of ethanol (50%, 70%, 85%, 96% ethanol) for dehydration.139 They were dried overnight and then mounted on a 30 mm diameter aluminum stub with an adhesive tape. The specimens were sputter coated with a 300 Armstrong gold coating in the Auto coater .The scanning electron micrographs were taken from SEM .Each specimen was scored blindly by two investigators specialized in Oral Biology. Six SEM photographs with different standardized magnifications were taken for each specimen which were later assessed using the indices, "Roughness and Loss of Tooth Substance Index" and "Smear Layer Index".17, 57 "Roughness and Loss of Tooth substance index" was analyzed taking the magnifications (×100, ×200, and × 500) into consideration. "Smear layer index" was analyzed using the magnifications (×1000, × 2000, and × 5000) into consideration. For computation of Root Roughness and Smear layer Index a single value was represented by taking mode of the three readings taken on three different magnifications of both indices. The micrographs were assessed by two examiners blinded to the treatment groups. Inter-examiner reliability was checked to ensure the calibration of the examiners by applying Intra-class Correlation Coefficient (ICC) test.

Data was analyzed using SPSS Version 21.Descriptive statistics was computed regarding patients age, gender, brushing and flossing habits. Similarly descriptive statistics regarding teeth were made using frequencies and percentages. Graphs were made like pie chart using frequencies and bar charts using means. Cross Tabulation was made between the test groups (Control, Gracey Curette, After five and Mini Five) versus "Roughness and Loss of Tooth substance Index". Similarly Cross Tabulation was made between the test groups versus "Smear Layer Index". Chi square test was applied to see the grade distribution among groups. P. value of 0.05 or less was considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Single Rooted Teeth diagnosed with severe chronic periodontitis
* Participants otherwise healthy
* Clinical Attachment Loss of >= 5mm
* Teeth with Millers Class 3 Mobility
* No alteration in root surface due to extraction procedure.

Exclusion Criteria:

* Teeth that had undergone root canal treatment
* Teeth associated with any periapical lesion
* History of scaling and root planing
* Any fractured teeth
* Any external resorption of root
* Any subgingival restoration or root caries

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2018-10-07 (Actual); Study Completion 2018-10-07 (Actual)

PRIMARY OUTCOMES:
Root Roughness | 1 week
  ROUGHNESS AND LOSS OF TOOTH SUBSTANCE INDEX
Smear Layer | 1 week
  Smear Layer Index

CONTACTS AND LOCATIONS:
Overall Officials: Sania Riaz, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dr Sania Riaz, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slot DE, Koster TJ, Paraskevas S, Van der Weijden GA. The effect of the Vector scaler system on human teeth: a systematic review. Int J Dent Hyg. 2008 Aug;6(3):154-65. doi: 10.1111/j.1601-5037.2008.00319.x. PMID 18768018
- [Background] Mittal A, Nichani AS, Venugopal R, Rajani V. The effect of various ultrasonic and hand instruments on the root surfaces of human single rooted teeth: A Planimetric and Profilometric study. J Indian Soc Periodontol. 2014 Nov-Dec;18(6):710-7. doi: 10.4103/0972-124X.147405. PMID 25624626
- [Background] Schwarz F, Aoki A, Sculean A, Georg T, Scherbaum W, Becker J. In vivo effects of an Er:YAG laser, an ultrasonic system and scaling and root planing on the biocompatibility of periodontally diseased root surfaces in cultures of human PDL fibroblasts. Lasers Surg Med. 2003;33(2):140-7. doi: 10.1002/lsm.10201. PMID 12913887
- [Background] Yaghini J, Naghsh N, Attaei E, Birang R, Birang E. Root Surface Roughness After Scaling and Root Planing with Er:YAG Laser Compared to Hand and Ultrasonic Instruments by Profilometry. J Dent (Tehran). 2015 Dec;12(12):899-905. PMID 27559349
- [Background] Dahiya P, Kamal R, Gupta R, Pandit N. Comparative evaluation of hand and power-driven instruments on root surface characteristics: A scanning electron microscopy study. Contemp Clin Dent. 2011 Apr;2(2):79-83. doi: 10.4103/0976-237X.83065. PMID 21957380
- [Background] Aspriello SD, Piemontese M, Levrini L, Sauro S. Ultramorphology of the root surface subsequent to hand-ultrasonic simultaneous instrumentation during non-surgical periodontal treatments: an in vitro study. J Appl Oral Sci. 2011 Jan-Feb;19(1):74-81. doi: 10.1590/s1678-77572011000100015. PMID 21437474
- [Derived] Riaz S, Ahmed S, Shabbir S, Khan ZR, Zaidi SJA, Naeem MM, Farooqui WA. Analysing root roughness and smear layer relationship by comparing contemporary dental curettes with conventional dental curettes: a randomised controlled trial. BMC Oral Health. 2022 Jun 17;22(1):237. doi: 10.1186/s12903-022-02268-1. PMID 35715802